CLINICAL TRIAL: NCT01609556
Title: A Phase 1, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of IMGN853 in Adults With Ovarian Cancer and Other FOLR1-Positive Solid Tumors
Brief Title: First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Mirvetuximab Soravtansine in Adults With Ovarian Cancer and Other Folate Receptor 1 (FOLR1)-Positive Solid Tumors
Acronym: IMGN853-0401
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMGN853-0401
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Tumors
Keywords: FOLR-1 solid tumors
MeSH Terms: conditions — Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine Q3W) (Experimental): Participants will receive mirvetuximab soravtansine intravenous (IV) infusion on Day 1 of every 21-day (every 3 weeks [Q3W]) cycle. Dose escalation for this group schedule will start at 0.15 milligrams per kilogram (mg/kg) and proceed through 7.0 mg/kg. Doses calculated initially based on participant's total body weight (TBW); then from protocol amendment 5 onwards, calculated based on adjusted ideal body weight (AIBW). Participants will continue to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever comes first, or until the sponsor terminate the study.
  Interventions: Drug: Mirvetuximab soravtansine
- Dose Escalation: Schedule B (Mirvetuximab Soravtansine Weekly) (Experimental): Participants will receive mirvetuximab soravtansine IV infusion on Days 1, 8, and 15 of every 28-day cycle. Dose escalation for this group schedule will start at 1.1 mg/kg (calculated based on AIBW) and proceed through 2.5 mg/kg. Participants will continue to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever comes first, or until the sponsor terminate the study.
  Interventions: Drug: Mirvetuximab soravtansine
- Dose Expansion:EOC Participants(Mirvetuximab Soravtansine Q3W) (Experimental): Participants with epithelial ovarian cancer (EOC) will receive mirvetuximab soravtansine 6.0 mg/kg (maximum tolerated dose [MTD]) IV infusion on Day 1 of every 21-day (Q3W) cycle (calculated based on AIBW). Participants will continue to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever comes first, or until the sponsor terminated the study.
  Interventions: Drug: Mirvetuximab soravtansine
- Dose Expansion: EC Participants(Mirvetuximab Soravtansine Q3W) (Experimental): Participants with endometrial cancer (EC) will receive mirvetuximab soravtansine 6.0 mg/kg (MTD) IV infusion on Day 1 of every 21-day (Q3W) cycle (calculated based on AIBW). Participants will continue to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever comes first, or until the sponsor terminate the study.
  Interventions: Drug: Mirvetuximab soravtansine

INTERVENTIONS:
Drug: Mirvetuximab soravtansine — Mirvetuximab soravtansine IV infusion will be administered as per dose and schedule specified in the respective arms.
  Other Names: IMGN853

SUMMARY:
The purpose of this study is to test mirvetuximab soravtansine (IMGN853) in participants with ovarian cancer and other FOLR-1 positive tumors.

DETAILED DESCRIPTION:
The study consists of a dose-escalation phase that will evaluate 2 dosing schedules (Schedule A and Schedule B) of mirvetuximab soravtansine and up to 5 dose-expansion groups at the maximum tolerated dose (MTD). The first 4 escalation cohorts will be single participant cohorts. Subsequent escalation cohorts will use a standard 3+3 design, with each cohort consisting of 3 or 4 to 6 participants. Data were collected and analysed for the escalation and expansion groups by dose schedule and not by individual dose.

ELIGIBILITY:
Inclusion Criteria

* Participants with advanced solid tumor that is refractory to standard treatment, for which no standard treatment is available, or the participant refuses standard therapy.
* Participants must be willing to provide an archival tumor tissue block or slides for biomarker analysis.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Time from prior therapy:

  1. Systemic anti-neoplastic therapy: five half-lives or four weeks, whichever is shorter (6 weeks for prior nitrosoureas or mitomycin C).
  2. Radiotherapy: wide-field radiotherapy (for example, greater than [>] 30 percent [%] of marrow-bearing bones) completed at least four weeks, or focal radiation completed at least two weeks, prior to starting study drug.
* Participants must have recovered or stabilized from all therapy-related toxicities.
* Major surgery (not including placement of vascular access device or tumor biopsies) must be completed four weeks prior to Day 1. Participants must have recovered or stabilized from the side effects prior to study treatment.
* Participants must have adequate hematologic, liver and kidney function.
* Participants with central nervous system (CNS) disease involvement are eligible if they have had brain metastases resected or have received radiation therapy ending at least 4 weeks prior to study day 1 and they meet all of the following criteria: Residual neurological symptoms less than or equal to (<=) Grade 1; No dexamethasone requirement; and Follow-up magnetic resonance imaging (MRI) shows no progression of treated lesions and no new lesions appearing.
* Participants must be willing and able to sign the informed consent form, and to adhere to the study visit schedule and other protocol requirements.
* Women of childbearing potential and men must agree to use effective contraceptive methods while on study and for at least twelve weeks after the last dose of study drug.
* Women of childbearing potential must have a negative pregnancy test prior to the first dose of study treatment.

Exclusion Criteria

* Grade >1 neuropathy.
* Any active or chronic corneal disorder, including, but not limited to the following: Sjogren's syndrome, Fuch's corneal dystrophy (requiring treatment), history of corneal transplantation, active herpetic keratitis, and also active ocular conditions requiring ongoing treatment/monitoring such as wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, presence of papilledema, acquired monocular vision.
* Serious concurrent illness, including, but not limited to the following:

  1. Clinically relevant active infection including known active hepatitis B or C, Human Immunodeficiency Virus (HIV) infection, varicella-zoster virus (shingles) or cytomegalovirus infection or any other known concurrent infectious disease, requiring IV antibiotics within 2 weeks of study enrollment.
  2. Significant cardiac disease such as recent myocardial infarction (<=6 months prior to Day 1), unstable angina pectoris, uncontrolled congestive heart failure (New York Heart Association >class II), uncontrolled hypertension (greater than or equal to [>=] Common Terminology Criteria for Adverse Events Version 4.03 [CTCAE v4.03] Grade 3), uncontrolled cardiac arrhythmias, severe aortic stenosis, or >=Grade 3 cardiac toxicity following prior chemotherapy.
  3. History of multiple sclerosis or other demyelinating disease, Eaton-Lambert syndrome (para-neoplastic syndrome), history of hemorrhagic or ischemic stroke within the last six months, or alcoholic liver disease.
  4. Previous clinical diagnosis of treatment-related pneumonitis.
* Any other concomitant anti-cancer treatment such as immunotherapy, biotherapy, radiotherapy, chemotherapy, investigative therapy, or high-dose steroids; however, low dose steroids and Luteinizing Hormone Releasing Hormone (LHRH) at doses that have been stable for >=14 days are permitted for participants with prostate cancer.
* Known hypersensitivity to previous monoclonal antibody therapy or maytansinoids.
* Prior history of solid tumor malignancy within the last 3 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer (participants must have shown no evidence of active disease for 2 years prior to enrollment).
* Concomitant administration of folate-containing vitamins.
* Participants who have received prior allogeneic or autologous bone marrow transplants.
* Women of childbearing potential who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2012-06-28 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - University of Kansas Medical Center Research Institute, Fairway, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - CTRC at the University of Texas Health Science Center, San Antonio, Texas
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 206 participants were enrolled in this study, of whom 69 participants (44 to receive Schedule A and 25 to receive Schedule B treatment) were entered in dose-escalation phase and 137 participants (113 with epithelial ovarian cancer [EOC] and 24 with endometrial cancer [EC]) were entered in dose-expansion phase. Doses calculated initially based on participant's total body weight (TBW); then from protocol amendment 5 onwards, calculated based on adjusted ideal body weight (AIBW).
Pre-assignment Details: Dose expansion Cohort 4 was planned to enroll relapsed/refractory non-small cell lung cancer (NSCLC) adenocarcinoma or bronchoalveolar carcinoma (BAC) but no participants were enrolled due to a company decision to focus on endometrial and ovarian carcinoma for the initial investigation.
Groups:
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W): Participants received mirvetuximab soravtansine 0.15 milligrams (mg)/kilogram (kg) intravenous (IV) infusion on Day 1 of every 21-day (every 3 weeks [Q3W]) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W): Participants received mirvetuximab soravtansine 0.5 mg/kg IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W): Participants received mirvetuximab soravtansine 1.0 mg/kg IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W): Participants received mirvetuximab soravtansine 2.0 mg/kg IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W): Participants received mirvetuximab soravtansine 3.3 mg/kg IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W): Participants received mirvetuximab soravtansine 5.0 mg/kg IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W): Participants received mirvetuximab soravtansine 6.0 mg/kg IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W): Participants received mirvetuximab soravtansine 7.0 mg/kg IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly): Participants received mirvetuximab soravtansine 1.1 mg/kg IV infusion on Days 1, 8, and 15 of every 28-day cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly): Participants received mirvetuximab soravtansine 1.8 mg/kg IV infusion on Days 1, 8, and 15 of every 28-day cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly): Participants received mirvetuximab soravtansine 2.0 mg/kg IV infusion on Days 1, 8, and 15 of every 28-day cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly): Participants received mirvetuximab soravtansine 2.5 mg/kg IV infusion on Days 1, 8, and 15 of every 28-day cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W): Participants with EOC, primary peritoneal cancer, or fallopian tube cancer resistant to platinum-based therapy received mirvetuximab soravtansine 6.0 mg/kg (maximum tolerated dose [MTD]) IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W): Participants with folate receptor 1 (FOLR1)-positive uterine cancer (that was advanced or recurrent and had received at least 1 platinum-based regimen, and no more than 5 prior systemic treatment regimens for EC) received mirvetuximab soravtansine 6.0 mg/kg (MTD) IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W): Participants with biopsy-accessible relapsed or refractory ovarian cancer, primary peritoneal cancer, or fallopian tube cancer received mirvetuximab soravtansine 6.0 mg/kg (MTD) IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W): Participants with EOC primary peritoneal cancer or fallopian tube cancer (that had relapsed following platinum-based therapy, excluding those participants with primary platinum refractory disease or low grade or clear cell ovarian cancer) received mirvetuximab soravtansine 6.0 mg/kg (MTD) IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
Period: Dose Escalation: Maximum 101.3 Weeks
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
Started | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 1 | 1 | 8 | 13 | 5 | 4 | 3 | 3 | 6 | 3 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Began New Anticancer Therapy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion: Maximum 124 Weeks
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46 | 24 | 27 | 40
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46 | 24 | 27 | 40
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 2
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 13 | 20 | 27
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 2
Not completed — Began New Anticancer Therapy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 5
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 3
Not completed — Other Than Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W): Participants received mirvetuximab soravtansine 0.15 mg/kg IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W): Participants with EOC, primary peritoneal cancer, or fallopian tube cancer resistant to platinum-based therapy received mirvetuximab soravtansine 6.0 mg/kg (MTD) IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W): Participants with FOLR1-positive uterine cancer (that was advanced or recurrent and had received at least 1 platinum-based regimen, and no more than 5 prior systemic treatment regimens for EC) received mirvetuximab soravtansine 6.0 mg/kg (MTD) IV infusion on Day 1 of every 21-day (Q3W) cycle. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W) | Total
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 46 | 24 | 27 | 40 | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 | 1 | 6 | 11 | 4 | 3 | 2 | 2 | 5 | 5 | 25 | 10 | 17 | 30 | 122
  >=65 years | 2 | 0 | 1 | 0 | 3 | 7 | 3 | 2 | 3 | 2 | 4 | 2 | 21 | 14 | 10 | 10 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 9 | 16 | 5 | 4 | 4 | 4 | 9 | 7 | 46 | 24 | 27 | 40 | 200
  Male | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 2 | 1 | 1 | 1 | 9 | 16 | 7 | 3 | 4 | 4 | 9 | 6 | 44 | 23 | 26 | 33 | 189
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 5
  White | 2 | 1 | 1 | 1 | 7 | 18 | 6 | 5 | 5 | 4 | 9 | 5 | 41 | 23 | 25 | 34 | 187
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Dose-Escalation Phase: Maximum Tolerated Dose (MTD) of Mirvetuximab Soravtansine
Description: MTD was defined as the highest dose at which 1 or fewer among 6 participants or less than or equal to (<=) 33 percent (%) experienced a dose-limiting toxicity (DLT) (calculated based on adjusted ideal body weight [AIBW]). AIBW was calculated as ideal body weight (IBW) + 0.4 * (actual weight - IBW), where IBW for men was 0.9 * height in centimeters (cm) - 88 and IBW for women was 0.9 * height in cm - 92. DLT was defined as a treatment-emergent adverse event (TEAE) or abnormal laboratory value related to study treatment (that is, assessed as unrelated to disease, intercurrent illness, or concomitant medications), including those TEAEs and abnormal laboratory values that resulted in a failure to meet the criteria for re-treatment.
Time Frame: Cycle 1 (21 days)
Population: Safety population included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: mg/kg
Groups:
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine Q3W): Participants received mirvetuximab soravtansine IV infusion on Day 1 of every 21-day (Q3W) cycle. Dose escalation started at 0.15 mg/kg and proceeded through 7.0 mg/kg. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule B (Mirvetuximab Soravtansine Weekly): Participants received mirvetuximab soravtansine IV infusion on Days 1, 8, and 15 of every 28-day cycle. Dose escalation started at 1.1 mg/kg and proceeded through 2.5 mg/kg. Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine Weekly)
Number analyzed (Participants) | 44 | 25
mg/kg | 6.0 | 2.0

2. Primary Outcome: Dose-Escalation Phase: Recommended Phase 2 Dose (RP2D) of Mirvetuximab Soravtansine
Description: RP2D was determined by MTD. MTD was defined as the highest dose at which 1 or fewer among 6 participants or <=33% experienced a DLT. DLT was defined as a TEAE or abnormal laboratory value related to study treatment (that is, assessed as unrelated to disease, intercurrent illness, or concomitant medications), including those TEAEs and abnormal laboratory values that resulted in a failure to meet the criteria for re-treatment. Available clinical data indicated that the MTD defined for the Q3W schedule was equal to the RP2D.
Time Frame: Cycle 1 (21 days)
Population: Safety population included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: mg/kg
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 44
mg/kg | 6.0

3. Secondary Outcome: Number of Participants With TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to study drug. Severity was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 on following scale: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening, Grade 5=death. Serious AEs include death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as any AE that emerged on or after the first dose, and within 28 days of the last dose.
Time Frame: From first dose of study drug up to 28 days after last dose of study drug (maximum exposure: 36 weeks for dose-escalation Schedule A, 101.3 weeks for dose-escalation Schedule B, 124 weeks for dose-expansion EOC, 33.3 weeks for dose-expansion EC)
Population: Safety population included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 46 | 24 | 27 | 40
Participants
  Any TEAE | 2 | 1 | 0 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 46 | 24 | 27 | 40
  SAEs | 2 | 1 | 0 | 0 | 0 | 5 | 1 | 2 | 2 | 3 | 4 | 4 | 18 | 11 | 9 | 17
  Grade >=3 TEAEs | 2 | 1 | 0 | 1 | 1 | 8 | 1 | 3 | 2 | 3 | 4 | 4 | 24 | 12 | 14 | 24

4. Secondary Outcome: Number of Participants With Shift From Baseline Grade <=2 in Clinical Laboratory Parameters to Grade 3 or Grade 4 on Study
Description: Laboratory parameters included serum chemistry (alanine aminotransferase [ALT]/serum glutamic pyruvic transaminase [SGPT], aspartate aminotransferase [AST]/serum glutamic oxaloacetic transaminase [SGOT], albumin, alkaline phosphatase, bilirubin, calcium, creatinine, glucose, magnesium, phosphorous, potassium, sodium), hematology (hemoglobin, lymphocytes, neutrophils, platelets, white blood cells) and coagulation (international normalized ratio [INR], partial thromboplastin time [PTT]). Clinically significant laboratory values were defined as per NCI CTCAE v.03 Grade 3 or higher. A grading (severity) scale was provided with grades ranging from 0 (none), 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening or disabling), to 5 (death). Only participants who shifted from a baseline value of Grade <=2 to a post-baseline Grade 3/4 on-treatment, are reported.
Time Frame: as for outcome 3
Population: Safety population included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 46 | 24 | 27 | 40
Participants
  Glucose: Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Magnesium: Grade 2 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  PTT: Grade 2 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Grade 0 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocytes: Grade 2 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination Findings and Vital Signs
Description: Physical examination included assessments of general appearance, skin, head (eyes, ears, nose, and throat), neck, lungs, heart, abdomen, back, lymph nodes, extremities, and neurological system. Vital signs included assessment of blood pressure, pulse rate, respiratory rate and body temperature.
Time Frame: as for outcome 3
Population: Safety population included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 46 | 24 | 27 | 40
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: Standard ECGs were performed in triplicate at 2- to 5-minute intervals during the study. A single ECG was performed at the end of treatment visit and as clinically indicated.
Time Frame: Baseline up to end of treatment (EOT) (up to maximum 124 weeks)
Population: Safety population included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 46 | 24 | 27 | 40
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0

7. Secondary Outcome: Number of Participants With Treatment-Emergent Ocular AEs
Description: Ocular AEs included keratopathy and blurred vision. An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to study drug. TEAEs were defined as any AE that emerged on or after the first dose, and within 28 days of the last dose.
Time Frame: as for outcome 3
Population: Safety population included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 46 | 24 | 27 | 40
Participants | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 5 | 0 | 3 | 0 | 2 | 24 | 9 | 14 | 18

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Mirvetuximab Soravtansine and Total M9346A Antibody at RP2D
Description: Pharmacokinetic (PK) parameters were calculated using standard non-compartmental methods. PK analysis of mirvetuximab soravtansine and total M9346A antibody is presented for a subgroup of participants who received 6.0 mg/kg (RP2D) mirvetuximab soravtansine at Cycle 1 and Cycle 3.
Time Frame: Cycle 1, 3: Day 1 (pre-infusion; within 10 minutes [min] of EOI; 2, 4, 6, 8 hrs post-infusion); Day 2, 3 (24, 48 hrs post-infusion); Day 4 or 5, 8, 15 (24 hrs post-infusion)
Population: PK Population included all participants who received at least 1 infusion of mirvetuximab soravtansine and had evaluable PK data. 'Overall number of participants analyzed' = participants who received mirvetuximab soravtansine at 6 mg/kg AIBW. 'Number analyzed' = participants evaluable for this outcome for specified categories.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Groups:
- Mirvetuximab Soravtansine 6.0 mg/kg AIBW: Participants received mirvetuximab soravtansine 6.0 mg/kg (calculated based on AIBW) on Day 1 of Cycle 1 and Cycle 3.
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
micrograms per milliliter (mcg/mL)
  Mirvetuximab soravtansine at Cycle 1 | 146.9 (30.14)
  Mirvetuximab soravtansine at Cycle 3: number analyzed (Participants) | 90
  Mirvetuximab soravtansine at Cycle 3 | 154.6 (33.08)
  Total M9346A antibody at Cycle 1 | 149.2 (33.74)
  Total M9346A antibody at Cycle 3: number analyzed (Participants) | 90
  Total M9346A antibody at Cycle 3 | 170.4 (40.55)

9. Secondary Outcome: Cmax of Free DM4 and S-Methyl DM4 at RP2D
Description: PK parameters were calculated using standard non-compartmental methods. PK analysis of free N2'-[4-[(3-carboxypropyl)dithio]-4-methyl-1-oxo-2-sulfopentyl]-N2'-deacetylmaytansine (DM4) and S-methyl DM4 is presented for a subgroup of participants who received 6.0 mg/kg (RP2D) mirvetuximab soravtansine at Cycle 1 and Cycle 3.
Time Frame: Cycle 1, 3: Day 1 (pre-infusion; within 10 min of EOI; 2, 4, 6, 8 hrs post-infusion); Day 2, 3 (24, 48 hrs post-infusion); Day 4 or 5, 8, 15 (24 hrs post-infusion)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
nanograms per milliliter (ng/mL)
  DM4 at Cycle 1: number analyzed (Participants) | 45
  DM4 at Cycle 1 | 5.014 (3.119)
  DM4 at Cycle 3: number analyzed (Participants) | 35
  DM4 at Cycle 3 | 5.016 (2.389)
  S-methyl DM4 at Cycle 1: number analyzed (Participants) | 45
  S-methyl DM4 at Cycle 1 | 12.43 (12.39)
  S-methyl DM4 at Cycle 3: number analyzed (Participants) | 35
  S-methyl DM4 at Cycle 3 | 9.974 (5.485)

10. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of Mirvetuximab Soravtansine and Total M9346A Antibody at RP2D
Description: PK parameters were calculated using standard non-compartmental methods. PK analysis of mirvetuximab soravtansine and total M9346A antibody is presented for a subgroup of participants who received 6.0 mg/kg (RP2D) mirvetuximab soravtansine at Cycle 1 and Cycle 3.
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours*milligrams/milliliter (hr*mg/mL)
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
hours*milligrams/milliliter (hr*mg/mL)
  Mirvetuximab soravtansine at Cycle 1 | 17.39 (4.341)
  Mirvetuximab soravtansine at Cycle 3: number analyzed (Participants) | 87
  Mirvetuximab soravtansine at Cycle 3 | 20.40 (5.144)
  Total M9346A antibody at Cycle 1 | 24.00 (7.316)
  Total M9346A antibody at Cycle 3: number analyzed (Participants) | 87
  Total M9346A antibody at Cycle 3 | 37.27 (12.54)

11. Secondary Outcome: AUC0-inf of Free DM4 and S-Methyl DM4 at RP2D
Description: PK parameters were calculated using standard non-compartmental methods. PK analysis of free DM4 and S-methyl DM4 is presented for a subgroup of participants who received 6.0 mg/kg (RP2D) mirvetuximab soravtansine at Cycle 1 and Cycle 3.
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours*nanograms/milliliter (hr*ng/mL)
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
hours*nanograms/milliliter (hr*ng/mL)
  DM4 at Cycle 1: number analyzed (Participants) | 38
  DM4 at Cycle 1 | 292.9 (129.2)
  DM4 at Cycle 3: number analyzed (Participants) | 27
  DM4 at Cycle 3 | 290.6 (98.52)
  S-methyl DM4 at Cycle 1: number analyzed (Participants) | 39
  S-methyl DM4 at Cycle 1 | 2656 (2722)
  S-methyl DM4 at Cycle 3: number analyzed (Participants) | 27
  S-methyl DM4 at Cycle 3 | 1928 (1108)

12. Secondary Outcome: Area Under the Plasma Concentration-Versus Time Curve From Time of Dose Until Tlast (AUClast) of Mirvetuximab Soravtansine and Total M9346A Antibody at RP2D
Description: as for outcome 10
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hr*mg/mL
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
hr*mg/mL
  Mirvetuximab soravtansine at Cycle 1 | 16.44 (4.177)
  Mirvetuximab soravtansine at Cycle 3: number analyzed (Participants) | 87
  Mirvetuximab soravtansine at Cycle 3 | 18.91 (4.940)
  Total M9346A antibody at Cycle 1 | 20.27 (5.903)
  Total M9346A antibody at Cycle 3: number analyzed (Participants) | 87
  Total M9346A antibody at Cycle 3 | 29.29 (9.613)

13. Secondary Outcome: AUClast of Free DM4 and S-Methyl DM4 at RP2D
Description: as for outcome 11
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
hr*ng/mL
  DM4 at Cycle 1: number analyzed (Participants) | 43
  DM4 at Cycle 1 | 246.0 (133.3)
  DM4 at Cycle 3: number analyzed (Participants) | 27
  DM4 at Cycle 3 | 270.1 (95.62)
  S-methyl DM4 at Cycle 1: number analyzed (Participants) | 45
  S-methyl DM4 at Cycle 1 | 2485 (2536)
  S-methyl DM4 at Cycle 3: number analyzed (Participants) | 27
  S-methyl DM4 at Cycle 3 | 1806 (1046)

14. Secondary Outcome: Terminal Half-Life (t1/2) of Mirvetuximab Soravtansine,Total M9346A Antibody, DM4, and S-Methyl DM4 at RP2D
Description: PK parameters were calculated using standard non-compartmental methods. PK analysis of mirvetuximab soravtansine, total M9346A antibody, DM4, and S-methyl DM4 is presented for a subgroup of participants who received 6.0 mg/kg (RP2D) mirvetuximab soravtansine at Cycle 1 and Cycle 3.
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
hours
  Mirvetuximab soravtansine at Cycle 1 | 119.4 (22.58)
  Mirvetuximab soravtansine at Cycle 3: number analyzed (Participants) | 90
  Mirvetuximab soravtansine at Cycle 3 | 127.8 (34.11)
  Total M9346A antibody at Cycle 1 | 186.7 (54.04)
  Total M9346A antibody at Cycle 3: number analyzed (Participants) | 90
  Total M9346A antibody at Cycle 3 | 218.8 (71.46)
  DM4 at Cycle 1: number analyzed (Participants) | 38
  DM4 at Cycle 1 | 73.80 (28.99)
  DM4 at Cycle 3: number analyzed (Participants) | 30
  DM4 at Cycle 3 | 80.62 (26.12)
  S-methyl DM4 at Cycle 1: number analyzed (Participants) | 39
  S-methyl DM4 at Cycle 1 | 122.2 (25.23)
  S-methyl DM4 at Cycle 3: number analyzed (Participants) | 32
  S-methyl DM4 at Cycle 3 | 130.4 (23.47)

15. Secondary Outcome: Clearance (CL) of Mirvetuximab Soravtansine and Total M9346A Antibody at RP2D
Description: as for outcome 10
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milliliters per hour (mL/hr)
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
milliliters per hour (mL/hr)
  Mirvetuximab soravtansine at Cycle 1: number analyzed (Participants) | 141
  Mirvetuximab soravtansine at Cycle 1 | 22.20 (6.476)
  Mirvetuximab soravtansine at Cycle 3: number analyzed (Participants) | 87
  Mirvetuximab soravtansine at Cycle 3 | 19.80 (4.953)
  Total M9346A antibody at Cycle 1: number analyzed (Participants) | 141
  Total M9346A antibody at Cycle 1 | 16.89 (7.155)
  Total M9346A antibody at Cycle 3: number analyzed (Participants) | 87
  Total M9346A antibody at Cycle 3 | 13.26 (4.956)

16. Secondary Outcome: CL of DM4 and S-Methyl DM4 at RP2D
Description: PK parameters were calculated using standard non-compartmental methods. PK analysis of DM4 and S-methyl DM4 is presented for a subgroup of participants who received 6.0 mg/kg (RP2D) mirvetuximab soravtansine at Cycle 1 and Cycle 3.
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liters per hour (L/hr)
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
Liters per hour (L/hr)
  DM4 at Cycle 1: number analyzed (Participants) | 38
  DM4 at Cycle 1 | 1421 (560.2)
  DM4 at Cycle 3: number analyzed (Participants) | 27
  DM4 at Cycle 3 | 1338 (438.8)
  S-methyl DM4 at Cycle 1: number analyzed (Participants) | 39
  S-methyl DM4 at Cycle 1 | 218.9 (128.5)
  S-methyl DM4 at Cycle 3: number analyzed (Participants) | 27
  S-methyl DM4 at Cycle 3 | 258.4 (173.8)

17. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Mirvetuximab Soravtansine, Free DM4, S-Methyl DM4, and Total M9346A Antibody at RP2D
Description: PK parameters were calculated using standard non-compartmental methods. PK analysis of mirvetuximab soravtansine, free DM4, S-methyl DM4, and total M9346A antibody is presented for a subgroup of participants who received 6.0 mg/kg (RP2D) mirvetuximab soravtansine at Cycle 1 and Cycle 3.
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
hours
  Mirvetuximab soravtansine at Cycle 1 | 3.80 [1.2 to 24]
  Mirvetuximab soravtansine at Cycle 3: number analyzed (Participants) | 90
  Mirvetuximab soravtansine at Cycle 3 | 3.20 [1.1 to 47]
  Total M9346A antibody at Cycle 1 | 3.60 [1.1 to 53]
  Total M9346A antibody at Cycle 3: number analyzed (Participants) | 90
  Total M9346A antibody at Cycle 3 | 3.20 [0.93 to 170]
  DM4 at Cycle 1: number analyzed (Participants) | 45
  DM4 at Cycle 1 | 5.80 [1.7 to 500]
  DM4 at Cycle 3: number analyzed (Participants) | 35
  DM4 at Cycle 3 | 5.00 [1.1 to 670]
  S-methyl DM4 at Cycle 1: number analyzed (Participants) | 45
  S-methyl DM4 at Cycle 1 | 49.0 [5.8 to 500]
  S-methyl DM4 at Cycle 3: number analyzed (Participants) | 35
  S-methyl DM4 at Cycle 3 | 23.0 [4.5 to 670]

18. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Mirvetuximab Soravtansine Free DM4, S-Methyl DM4, and Total M9346A Antibody at RP2D
Description: as for outcome 17
Time Frame: as for outcome 9
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Mirvetuximab Soravtansine 6.0 mg/kg AIBW
Number analyzed (Participants) | 142
Liters
  Mirvetuximab soravtansine at Cycle 1: number analyzed (Participants) | 141
  Mirvetuximab soravtansine at Cycle 1 | 3.198 (0.7422)
  Mirvetuximab soravtansine at Cycle 3: number analyzed (Participants) | 87
  Mirvetuximab soravtansine at Cycle 3 | 3.172 (1.022)
  Total M9346A antibody at Cycle 1: number analyzed (Participants) | 141
  Total M9346A antibody at Cycle 1 | 3.744 (0.9183)
  Total M9346A antibody at Cycle 3: number analyzed (Participants) | 87
  Total M9346A antibody at Cycle 3 | 3.671 (1.185)
  DM4 at Cycle 1: number analyzed (Participants) | 38
  DM4 at Cycle 1 | 107400 (38770)
  DM4 at Cycle 3: number analyzed (Participants) | 27
  DM4 at Cycle 3 | 114300 (48740)
  S-methyl DM4 at Cycle 1: number analyzed (Participants) | 39
  S-methyl DM4 at Cycle 1 | 41590 (27890)
  S-methyl DM4 at Cycle 3: number analyzed (Participants) | 27
  S-methyl DM4 at Cycle 3 | 47520 (40440)

19. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With Objective Response as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: ORR was defined as percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). CR: Disappearance of all target or non-target lesions. All pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR: At least 30 percent (%) decrease in the sum of the longest diameters (SoD) of target lesions, taking as reference the baseline SoD.
Time Frame: From first dose of study drug until first BOR of CR or PR (maximum exposure: 36 weeks for dose-escalation Schedule A, 101.3 weeks for dose-escalation Schedule B, 124 weeks for dose-expansion EOC, 33.3 weeks for dose-expansion EC)
Population: Efficacy-evaluable population included participants who had radiographic assessment at baseline, received at least 1 dose of study drug, and had at least 1 post-dose tumor assessment or died or clinically progressed within 105 days of last dose. Data was only collected and reported combined for dose-escalation phase and not by individual doses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Escalation: Schedule A (Mirvetuximab Soravtansine Q3W): Participants received mirvetuximab soravtansine IV infusion on Day 1 of every 21-day (Q3W) cycle. Dose escalation started at 0.15 mg/kg and proceeded through 7.0 mg/kg. Doses calculated initially based on participant's TBW; then from protocol amendment 5 onwards, calculated based on AIBW. The doses evaluated during dose escalation for Schedule A, TBW were: 0.15 mg/kg (n=2); 0.5 mg/kg; 1.0 mg/kg, and 2.0 mg/kg (n=1, in each); 3.3 mg/kg (n=9); 5.0 mg/kg (n=11); and 7.0 mg/kg (n=5). The doses evaluated during dose escalation for Schedule A, AIBW were: 5.0 mg/kg (n=7); and 6 mg/kg (n=7). Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Escalation: Schedule B (Mirvetuximab Soravtansine Weekly): Participants received mirvetuximab soravtansine IV infusion on Days 1, 8, and 15 of every 28-day cycle. Dose escalation started at 1.1 mg/kg and proceeded through 2.5 mg/kg (calculated based on AIBW). The doses evaluated during dose escalation for Schedule B, AIBW were: 1.1 mg/kg (n=5); 1.8 mg/kg (n=4), 2.0 mg/kg (n=9); and 2.5 mg/kg (n=7). Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Expansion:EOC Participants(Mirvetuximab Soravtansine Q3W): Participants with EOC received mirvetuximab soravtansine 6.0 mg/kg (MTD) IV infusion on Day 1 of every 21-day (Q3W) cycle (calculated based on AIBW). Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
- Dose Expansion: EC Participants(Mirvetuximab Soravtansine Q3W): Participants with EC received mirvetuximab soravtansine 6.0 mg/kg (MTD) IV infusion on Day 1 of every 21-day (Q3W) cycle (calculated based on AIBW). Participants continued to receive mirvetuximab soravtansine (for clinical benefit) until unacceptable toxicity or withdrawal of consent, whichever came first, or until the sponsor terminated the study.
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine Weekly) | Dose Expansion:EOC Participants(Mirvetuximab Soravtansine Q3W) | Dose Expansion: EC Participants(Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 43 | 24 | 113 | 24
percentage of participants | 5 [0.6 to 15.8] | 13 [2.7 to 32.4] | 30 [21.8 to 39.4] | 8 [1.0 to 27.0]

20. Secondary Outcome: Duration of Response (DOR) as Assessed by RECIST v1.1
Description: DOR was defined as the time from the date of the first response (CR or PR), whichever was recorded first, until the date of progressive disease (PD). PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase. DOR was only defined for participants who had a BOR of CR or PR using the method of Kaplan-Meier.
Time Frame: From the date of first response (CR or PR) until the date of PD (maximum exposure: 36 weeks for dose-escalation Schedule A, 101.3 weeks for dose-escalation Schedule B, 124 weeks for dose-expansion EOC, 33.3 weeks for dose-expansion EC)
Population: Efficacy-evaluable population included participants who had radiographic assessment at baseline, received at least 1 dose of study drug, and had at least 1 post-dose tumor assessment or died or clinically progressed within 105 days of last dose. 'Overall number of participants analyzed'=participants who had a BOR of CR or PR. Data by group only.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine Weekly) | Dose Expansion:EOC Participants(Mirvetuximab Soravtansine Q3W) | Dose Expansion: EC Participants(Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 2 | 3 | 34 | 2
weeks | 21.3 [18.4 to 24.1] | 60.2 [44.3 to 76.1] | 19.3 [18.0 to 34.0] | 28.6 [NA to NA] — Due to smaller number of events, 95% CI could not be calculated.

21. Secondary Outcome: Progression-Free Survival (PFS) as Assessed by RECIST v1.1
Description: PFS was defined as the time from initiation of study drug until PD or death whichever occurred first, estimated using the Kaplan-Meier method. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions and appearance of new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: From first dose of study drug until PD or death whichever occurred first (maximum exposure: 36 weeks for dose-escalation Schedule A, 101.3 weeks for dose-escalation Schedule B, 124 weeks for dose-expansion EOC, 33.3 weeks for dose-expansion EC)
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine Weekly) | Dose Expansion:EOC Participants(Mirvetuximab Soravtansine Q3W) | Dose Expansion: EC Participants(Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 43 | 24 | 113 | 24
months | 2.6 [1.3 to 3.3] | 3.9 [1.8 to 11.1] | 4.3 [3.9 to 5.4] | 2.8 [1.2 to 4.2]

22. Secondary Outcome: Time to Progression (TTP) as Assessed by RECIST v1.1
Description: TTP was defined as the time from initiation of study drug until PD, estimated using the method of Kaplan-Meier. PD: At least a 20% increase in the SoD of target lesion, taken as reference the smallest (nadir) SoD since and including baseline. In addition to the relative increase of 20%, the SoD must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of non-target lesions and appearance of new lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: From first dose of study drug until PD (maximum exposure: 36 weeks for dose-escalation Schedule A, 101.3 weeks for dose-escalation Schedule B, 124 weeks for dose-expansion EOC, 33.3 weeks for dose-expansion EC)
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine Weekly) | Dose Expansion:EOC Participants(Mirvetuximab Soravtansine Q3W) | Dose Expansion: EC Participants(Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 43 | 24 | 113 | 24
months | 2.7 [1.3 to 3.3] | 3.9 [1.8 to 11.1] | 4.4 [4.0 to 5.6] | 2.8 [1.2 to 6.9]

23. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA)
Description: During the conduct of the study, a single immunogenicity assay was developed to concurrently detect human antibodies against all components of mirvetuximab soravtansine, including the humanized anti-FOLR1 antibody, the cleavable disulfide linker, and the cytotoxic maytansinoid, DM4. Therefore, immunogenicity results were reported as ADA titers, and did not distinguish between human anti-drug or anti-human titers.
Time Frame: Baseline up to follow-up visit (maximum exposure: 36 weeks for dose-escalation Schedule A, 101.3 weeks for dose-escalation Schedule B, 124 weeks for dose-expansion EOC, 33.3 weeks for dose-expansion EC)
Population: Immunogenicity population included all participants who received at least 1 infusion of mirvetuximab soravtansine and had evaluable immunogenicity data.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 9 | 18 | 7 | 5 | 5 | 4 | 9 | 7 | 46 | 24 | 27 | 40
Participants | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 2 | 2

24. Secondary Outcome: Number of Participants With Gynecologic Cancer Intergroup (GCIG) CA-125 Criteria Clinical Responses
Description: CA-125 response was defined as at least 50% reduction in CA-125 levels from baseline. The date of response corresponded to the date when the CA 125 level was first reduced by 50%.
Time Frame: From first dose of study drug until CA-125 response (maximum exposure: 36 weeks for dose-escalation Schedule A, 101.3 weeks for dose-escalation Schedule B, 124 weeks for dose-expansion EOC, 33.3 weeks for dose-expansion EC)
Population: CA-125 evaluable population included participants who had a baseline CA-125 value greater than or equal to (>=) 2 * upper limit of normal (ULN), received at least 1 dose of study drug, and had at least 1 post-dose CA-125 assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 3 | 10 | 2 | 3 | 2 | 2 | 4 | 5 | 31 | 12 | 20 | 26
Participants | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 2 | 2 | 3 | 23 | 4 | 11 | 17

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days after last dose of study drug (maximum exposure: 36 weeks for dose-escalation Schedule A, 101.3 weeks for dose-escalation Schedule B, 124 weeks for dose-expansion EOC, 33.3 weeks for dose-expansion EC)
Description: Safety population included all participants who were enrolled and received at least 1 dose of study drug. AEs (serious and non-serious) and deaths occurred during TEAE period were reported. Data was only collected and reported by combined groups for the dose-escalation phase and not by individual doses.
Arm/Group | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W)
All-Cause Mortality (participants affected / at risk) | 2/2 | 0/1 | 0/1 | 0/1 | 0/9 | 1/18 | 0/7 | 0/5 | 0/5 | 0/4 | 1/9 | 0/7 | 4/46 | 4/24 | 1/27 | 4/40
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/1 | 1/1 | 0/1 | 0/9 | 5/18 | 1/7 | 2/5 | 2/5 | 3/4 | 4/9 | 4/7 | 18/46 | 11/24 | 9/27 | 17/40
Other Adverse Events (participants affected / at risk) | 2/2 | 0/1 | 1/1 | 1/1 | 9/9 | 18/18 | 7/7 | 5/5 | 5/5 | 4/4 | 9/9 | 7/7 | 45/46 | 24/24 | 27/27 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) (N=2) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) (N=1) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) (N=1) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) (N=1) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) (N=9) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) (N=18) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) (N=7) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) (N=5) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) (N=5) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) (N=4) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) (N=9) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) (N=7) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) (N=46) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) (N=24) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) (N=27) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W) (N=40)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 7
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal opacity (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 4 | 7
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.15 mg/kg Q3W) (N=2) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 0.5 mg/kg Q3W) (N=1) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 1.0 mg/kg Q3W) (N=1) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 2.0 mg/kg Q3W) (N=1) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 3.3 mg/kg Q3W) (N=9) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 5.0 mg/kg Q3W) (N=18) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 6.0 mg/kg Q3W) (N=7) | Dose Escalation: Schedule A (Mirvetuximab Soravtansine 7.0 mg/kg Q3W) (N=5) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.1 mg/kg Weekly) (N=5) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 1.8 mg/kg Weekly) (N=4) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.0 mg/kg Weekly) (N=9) | Dose Escalation: Schedule B (Mirvetuximab Soravtansine 2.5 mg/kg Weekly) (N=7) | Dose Expansion: Cohort 1 (Mirvetuximab Soravtansine Q3W) (N=46) | Dose Expansion: Cohort 2 (Mirvetuximab Soravtansine Q3W) (N=24) | Dose Expansion: Cohort 3 (Mirvetuximab Soravtansine Q3W) (N=27) | Dose Expansion: Cohort 5 (Mirvetuximab Soravtansine Q3W) (N=40)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 7 | 2 | 2 | 2 | 1 | 5 | 3 | 24 | 8 | 10 | 23
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 4 | 1 | 2 | 3 | 2 | 6 | 3 | 19 | 10 | 9 | 19
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 5 | 1 | 0 | 0 | 1 | 3 | 1 | 4 | 2 | 4 | 7
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 2 | 2 | 3 | 2 | 15 | 5 | 6 | 10
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 2 | 2 | 9 | 7 | 8 | 10
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 5 | 0 | 3 | 0 | 2 | 23 | 7 | 11 | 16
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 2
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 8 | 1 | 2 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal pigmentation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 2 | 1 | 3 | 1 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 3 | 0 | 7 | 2 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 2 | 4 | 4 | 3 | 1 | 1 | 4 | 3 | 19 | 12 | 12 | 23
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 6 | 3 | 1 | 4
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 4 | 2 | 1 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 4 | 1 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 5
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 4 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 9 | 8 | 5 | 15
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 7 | 8 | 3 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 10 | 6 | 1 | 8
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 2 | 3 | 1 | 5 | 6 | 9 | 6 | 6 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 3 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 9 | 2 | 2 | 7
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 6 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 2
Facial neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 2 | 0 | 1 | 0 | 2 | 7 | 3 | 7 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 2 | 0 | 1 | 0 | 2 | 9 | 5 | 8 | 11
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 4 | 5 | 1 | 5
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 1 | 3 | 8 | 2 | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 5 | 2 | 5 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 5
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 3 | 1 | 6 | 2 | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 7 | 3 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sweating fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 9 | 3 | 2 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 4 | 2 | 1 | 4
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 3 | 1 | 1 | 8
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 3 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 7 | 4 | 5 | 9
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 1 | 3 | 6
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal deposits (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 6 | 6
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 6 | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 2 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 3
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thyroid pain (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 5
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site discolouration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Necrosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 3 | 5
Corneal epithelial microcysts (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 2
Corneal cyst (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1
Corneal disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vitreous degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal lesion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation decreased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lagophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Posterior capsule opacification (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous adhesions (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperreflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal stoma output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Waist circumference increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomal hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arterial intramural haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Perineal rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Right ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limbal stem cell deficiency (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-09-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT01609556/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT01609556/SAP_001.pdf